CLINICAL TRIAL: NCT05512377
Title: Brightline-2: A Phase IIa/IIb, Open-label, Single-arm, Multi-centre Trial of BI 907828 (Brigimadlin) for Treatment of Patients With Locally Advanced / Metastatic, MDM2 Amplified, TP53 Wild-type Biliary Tract Adenocarcinoma, Pancreatic Ductal Adenocarcinoma, or Other Selected Solid Tumours
Brief Title: Brightline-2: A Study to Test Whether Brigimadlin (BI 907828) Helps People With Cancer in the Biliary Tract, Pancreas, Lung or Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1403-0011; 2023-506369-79-00 (Other: CTIS); U1111-1292-3392 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP)); 2022-001500-18 (EudraCT Number)
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Neoplasms; Solid Tumors; Biliary Tract Cancer; Lung Neoplasms; Bladder Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms | interventions — brigimadlin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- brigimadlin (BI 907828) treatment arm (Experimental)
  Interventions: Drug: brigimadlin

INTERVENTIONS:
Drug: brigimadlin — brigimadlin
  Other Names: BI 907828

SUMMARY:
This study is open to adults with advanced cancer in the biliary tract, pancreas, lung, or bladder. This is a study for people for whom previous treatment was not successful or no treatment exists.

The purpose of this study is to find out whether a medicine called BI 907828 helps people with cancer in the biliary tract, pancreas, lung, or bladder. BI 907828 is a so-called MDM2 inhibitor that is being developed to treat cancer. All participants take BI 907828 as a tablet once every 3 weeks. Participants may continue to take BI 907828 as long as they benefit from treatment and can tolerate it. They visit the study site regularly. At the study site, doctors regularly check the size of the tumour and whether it has spread to other parts of the body. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a solid tumour which meets the criteria for an open trial cohort:

  * Cohorts 1 and 1-CN (biliary tract adenocarcinoma): Locally advanced or metastatic biliary tract adenocarcinoma (intra- and extrahepatic cholangiocarcinoma, gallbladder cancer, and ampullary cancer).Patients must have unresectable disease and have received all available conventional therapies known to confer clinical benefit for their disease based on local approved standards; or (in the opinion of the investigator) patients are unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy.
  * Cohort 2 (pancreatic ductal adenocarcinoma): Locally advanced or metastatic pancreatic ductal adenocarcinoma. Patients must have unresectable disease and have received all available conventional therapies known to confer clinical benefit for their disease based on local approved standards.
  * Cohort 3 (lung adenocarcinoma): Locally advanced or metastatic lung adenocarcinoma. Patients must have unresectable disease and have received all available conventional therapies known to confer clinical benefit for their disease based on local approved standards.
  * Cohort 4 (urothelial bladder cancer): Locally advanced or metastatic urothelial bladder cancer. Patients must have unresectable disease and have received all available conventional therapies known to confer clinical benefit for their disease based on local approved standards.
* Written pathology report / molecular profiling report indicating Mouse double minute 2 homolog (MDM2) amplification or a copy number ≥8 and tumor protein 53 (TP53) wild-type status. This must have been confirmed with a tissue-based test. A test with liquid biopsy is not accepted.
* Archival tissue (formalin fixed paraffin embedded [FFPE] tumour blocks or slides) must be provided for retrospective confirmation of MDM2 amplification and TP53 status.
* Presence of at least 1 measurable target lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Patient must be willing to donate mandatory blood samples for the pharmacokinetics, pharmacodynamics, and biomarker analyses
* Adequate organ function
* All toxicities related to previous anti-cancer therapies have resolved to ≤Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 prior to trial treatment administration (except for alopecia and amenorrhea / menstrual disorders which can be of any grade and peripheral neuropathy which must be ≤CTCAE Grade 2).
* Life expectancy ≥3 months at the start of treatment in the opinion of the investigator.
* Provision of signed and dated, written informed consent form (ICF) in accordance with ICH-GCP and local legislation prior to any trial-specific procedures, sampling, or analyses.
* Male or female patients ≥18 years old at the time of signature of the ICF. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use 2 medically acceptable methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at screening, during trial participation, and until 6 months and 12 days after last dose for women and 102 days after last dose for men. A list of contraception methods meeting these criteria is provided in the patient information.

Exclusion Criteria:

* Previous administration of brigimadlin (BI 907828) or any other MDM2-p53 or mouse double minute 4 (MDMX, MDM4)-p53 antagonist.
* Active bleeding, significant risk of haemorrhage (e.g. previous severe gastrointestinal bleeding, previous haemorrhagic stroke at any time), or current bleeding disorder (e.g. haemophilia, von Willebrand disease).
* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to start of trial treatment or planned within 6 months after screening (e.g. hip replacement).
* Clinically significant previous or concomitant malignancies in the opinion of the investigator affecting the efficacy and/or outcome of the trial.
* Patients who must or intend to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Currently enrolled in another investigational device or drug trial.
* Any history of, or concomitant condition that, in the opinion of the investigator, would compromise the patient's ability to comply with the trial or interfere with the evaluation of the safety and efficacy of the trial drug.
* Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the patient an unreliable trial participant).

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Objective response (OR) | Up to 30 months
  OR is defined as a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.1.

SECONDARY OUTCOMES:
Duration of objective response (DOR) | Up to 30 months
  DOR is defined as the time from first documented confirmed objective response (OR) until the earliest date of disease progression or death among patients with confirmed objective response.
Progression-free survival (PFS) | Up to 30 months
  PFS is defined as the time from treatment start until the earliest date of tumour progression according to RECIST version 1.1 or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 50 months
  OS is defined as the time from treatment start until death from any cause.
Disease control (DC) | Up to 30 months
  DC is defined as a best overall response of CR, PR, or stable disease (SD) where best overall response is defined according to RECIST version 1.1.
Occurrence of treatment-emergent adverse events (AEs) during the on-treatment period | Up to 30 months
Occurrence of treatment-emergent AEs leading to trial drug discontinuation during the on-treatment period | Up to 30 months
Change from baseline in European Organisation for Research and Treatment (EORTC) Quality of Life Questionnaire (QLQ)-C30 physical functioning domain score | Up to 30 months
  The QLQ-C30 comprises 30 questions. The QLQ-C30 incorporates both multi-items scales and single-item measures. These include 1 global health status/QoL scale, 5 functional scales, 3 symptoms scales and 6 single items to assess dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function, symptoms and financial difficulties and 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life.
Change from baseline in EORTC QLQ-C30 fatigue domain score | Up to 30 months
  It is part of QLQ-C30 and uses 4-point scale (1=not at all to 4=very much)
Change from baseline in EORTC QLQ-C30 role functioning domain score | Up to 30 months
  It is part of QLQ-C30 and uses 4-point scale (1=not at all to 4=very much)
Change from baseline in EORTC QLQ-BIL21 tiredness domain score | Up to 30 months
  The QLQ-BIL21 is specific for the assessment of quality of life in patients with cholangiocarcinoma and cancer of the gallbladder. It consists of 21 questions with a 4-point scale (1=not at all to 4=very much), and the tiredness domain is part of it.

CONTACTS AND LOCATIONS:
Locations (60):
- United States (18):
  - Southern Cancer Center, Mobile, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Providence Medical Foundation-Santa Rosa -69764, Santa Rosa, California
  - Rocky Mountain Cancer Centers-Lone Tree-69498, Lone Tree, Colorado
  - Johns Hopkins Sidney Kimmel Cancer Center at Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - University of Michigan Health System, Ann Arbor, Michigan
  - Nebraska Cancer Specialists-Omaha-69066, Omaha, Nebraska
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oncology Associates of Oregon, PC, Eugene, Oregon
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Prince of Wales Hospital-Randwick-66496, Randwick, New South Wales
  - ICON-South Brisbane-69267, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Austin Health, Heidelberg, Victoria
- Austria (2):
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
  - LK Wiener Neustadt, Wiener Neustadt
- Belgium (2):
  - Edegem - UNIV UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- France (2):
  - CTR Georges-François Leclerc, Dijon
  - INS Gustave Roussy, Villejuif
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Krankenhaus Nordwest, Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum der Universität München AÖR, München
  - Universitätsklinikum Ulm, Ulm
- Japan (7):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Kanagawa Cancer Center, Kanagawa, Yokohama
  - Tohoku University Hospital, Miyagi, Sendai
  - Osaka International Cancer Institute, Osaka, Osaka
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
  - Yamaguchi University Hospital, Yamaguchi, Ube
- King Abdul Aziz Medical City, Riyadh, Saudi Arabia
- National University Hospital-Singapore-42005, Singapore, Singapore
- Rainbow Oncology, KwaZulu, South Africa
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (2):
  - University Hospital Bern, Bern
  - University Hospital Geneva, Geneva
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (2):
  - Songklanagarind Hospital, Hat Yai
  - Srinagarind Hospital, Muang
- University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Yoo C, Lamarca A, Choi HJ, Vogel A, Pishvaian MJ, Goyal L, Ueno M, Marten A, Teufel M, Geng L, Morizane C. Brightline-2: a phase IIa/IIb trial of brigimadlin (BI 907828) in advanced biliary tract cancer, pancreatic ductal adenocarcinoma or other solid tumors. Future Oncol. 2024;20(16):1069-1077. doi: 10.2217/fon-2023-0963. Epub 2024 Jan 12. PMID 38214149
- See also: Related Info — http://www.mystudywindow.com